CLINICAL TRIAL: NCT02140723
Title: PART1 - a Prospective Phase II Study to Evaluate the Impact of TP53 Gene Mutations in Patients With Preoperative Radiotherapy for T2 and T3 Rectal Cancer
Brief Title: p53 and Response to Preoperative Radiotherapy for T2 and T3
Acronym: PART1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniela Kandioler, Unif. Prof. Dr., Medical University of Vienna
Other Study IDs: PART1
Record Dates: First submitted 2014-04-30; First posted 2014-05-16 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Rectal Cancer
Keywords: preoperative short course radiotherapy; delay of surgery; rectal cancer; TP53; predictive marker; MRT imaging
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood diagnostic tumor biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- preoperative short course radiation: preoperative short course radiation with 8 weeks delay of surgery
  Interventions: Radiation: preoperative short course radiation

INTERVENTIONS:
Radiation: preoperative short course radiation

SUMMARY:
Background:

Meta-analyses of large randomized trials proved the superiority of preoperative short course radiation and surgery, as compared with surgery alone. Short course radiation results in a 50% reduction in terms of local relapse in stage II and III rectal cancer patients. Patients with complete pathological remission additionally show a significant survival benefit. Complete pathological remission (pCR) occurs in 8% after preoperative radiation and in >16% if the interval between radiation and surgery is at least 8 weeks.

It is generally accepted that mutations in the TP53 gene represent a crucial defect in the apoptosis pathway. Radiation therapy is suggested to act via induction of apoptosis in irradiated cells. Therefore, it is expected that a defect in the TP53 gene has an effect on the success of radiation therapy.

Currently available imaging tools are hardly able to diagnose response to radiation therapy correctly, as this does not essentially correlate with tumor size.

Method:

Aim of this prospective observation study is to strengthen the hypothesis that the TP53 genotype is a promising marker to predict response to radiation therapy in rectal cancer patients. Consequently, the expected results will justify prospective, randomized intervention trials to obtain level of evidence I for the p53 marker hypothesis. Trial endpoint is downstaging and pCR rate. Tumor stage and pathological remission will be evaluated by MRT and pathohistology and correlated to the TP53 genotype of the diagnostic biopsy. Additionally, we will investigate the applicability of novel imaging modalities in magnet resonance tomography to monitor response to radiotherapy.

The objective of this study is

* to evaluate the effect of a genetic tumor marker (TP53 genotype) on the response to preoperative short course radiation (in terms of downstaging and pCR rate)
* to evaluate the applicability of novel magnet resonance tomography imaging modalities to monitor response to preoperative short time radiation.

Conclusion:

The prospective evaluation of the potential predictive marker TP53 may bring us one-step closer to an individualized therapy regimen, which allows the restriction of preoperative radiation in rectal cancer to those patients who will benefit.

ELIGIBILITY:
Inclusion Criteria:

Patients who are eligible for this observational study will be treated according to current standards with preoperative short course radiation (5x5 Gy) and a subsequent interval to surgery of at least 8 to maximum 16 weeks.

According to standards of rectal cancer therapy, eligible patients will meet the following criteria:

* Histologically confirmed adenocarcinoma of the rectum
* Tumor staging with MRI
* Inferior margin of the tumor located not farther than 15 cm from anal verge and below the level of S1-2
* Tumor stage T2 and T3
* No evidence of metastatic disease
* No prior tumor therapy for rectal or pelvic cancers (surgery, radio-, chemo-, immunotherapy, molecular target therapy, or any other type of tumor therapy)
* Medical fitness of the patient for treatment (decided by the involved physician)
* Patient compliance
* Signed informed consent from the patient or a legal representative, for the analysis of the tumor including genetic analyses of the tumor DNA.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons

* Clinical stage T1 (appropriate for local excision),
* Clinical stage T4 (Radio/Chemotherapy)
* Clinical stage M+ (distant metastases)
* No tumor staging with MRI
* Inoperability (technical or functional)
* Prior tumor therapy of the pelvis
* Concurrent administration of any other tumor therapy
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Serious concomitant disorders or attitudes of the patient that would compromise the safety of the patient or his/her ability to complete the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients with clinical staging T2/T3 Nx M0
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Interaction between the status of the biomarker TP53 and response to treatment | weeks 12-16 after treatment
  Primary outcome measure is the interaction between the status of the biomarker TP53 and response to radiation.
  The TP53 maker status is determined by standardized gene specific sequencing of the TP53 using DNA from formalin fixed paraffin embedded material from diagnostic biopsies.
  Response to treatment is determined by "down sizing" - down sizing will be measured by comparison of pretreatment T stage with pathohistological post treatment T stage . Pretreatement T stage is assessed with MRI, and supported by endosonography. Posttreatment T stage will be assessed prior to operation with MRI and after resection in the pathohistological specimen. The postreatment MRI results will be compared pathohistology.

SECONDARY OUTCOMES:
pCR rate | 12-16 weeks after treatment
  pCR - pathohistological complete resmission as assessed in surgical specimen
complete resection rate | 12-16 weeks after treatment
  Patholohistological assessment
relapse | 3 years
  local and distant relapse
overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Kandioler, MD, Study Chair — MUW
Locations (1):
- Medical University of Vienna, Department of Surgery, Vienna, Austria

REFERENCES:
- [Background] Kandioler D, Zwrtek R, Ludwig C, Janschek E, Ploner M, Hofbauer F, Kuhrer I, Kappel S, Wrba F, Horvath M, Karner J, Renner K, Bergmann M, Karner-Hanusch J, Potter R, Jakesz R, Teleky B, Herbst F. TP53 genotype but not p53 immunohistochemical result predicts response to preoperative short-term radiotherapy in rectal cancer. Ann Surg. 2002 Apr;235(4):493-8. doi: 10.1097/00000658-200204000-00006. PMID 11923604
- See also: Homepage of the p53-research group — http://www.p53.at